CLINICAL TRIAL: NCT03339752
Title: A Single-center, Open-label, One-sequence, Two-treatment Study to Investigate the Effect of ACT-541468 at Steady State on the Pharmacokinetics of Rosuvastatin in Healthy Male Subjects
Brief Title: A Study in Healthy Male Subjects to Investigate Whether Administration of ACT-541468 Can Affect the Fate in the Body (Amount and Time of Presence in the Blood) of Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ID-078-106
Record Dates: First submitted 2017-10-26; First posted 2017-11-13 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Rosuvastatin Calcium; daridorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): Rosuvastatin Day 1
  Interventions: Drug: Rosuvastatin
- Treatment B1 (Experimental): ACT-541468 Day 5 to Day 7
  Interventions: Drug: ACT-541468
- Treatment B2 (Other): Rosuvastatin Day 8; ACT-541468 Day 8 to Day 12
  Interventions: Drug: Rosuvastatin; Drug: ACT-541468

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg tablet
  Arms: Treatment A; Treatment B2
Drug: ACT-541468 — 25 mg hard capsule
  Arms: Treatment B1; Treatment B2

SUMMARY:
A study in healthy male subjects to investigate whether administration of ACT-541468 can affect the fate in the body (amount and time of presence in the blood) of rosuvastatin

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study mandated procedure;
* Healthy male subjects aged 18 to 45 years (inclusive) at screening;
* Body mass index of 18.0 to 28.0 kg/m2 (inclusive) at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to ACT-541468, rosuvastatin, any drug of the same classes, or any of their excipients;
* Any contraindication for rosuvastatin treatment;
* History or clinical evidence of myopathy;
* Asian or Indian-Asian ethnicity;
* Known hypersensitivity or allergy to natural rubber latex;
* Previous exposure to ACT-541468;
* Treatment with rosuvastatin within 3 months prior to screening;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Effect of ACT-541468 at steady-state on Cmax of single-dose rosuvastatin | During administration of rosuvastatin (Treatment A) and both rosuvastatin and ACT-541468 (Treatment B2); i.e. for about 2 weeks.
  Effect of ACT-541468 at steady-state on Cmax of single-dose rosuvastatin
Effect of ACT-541468 at steady-state on tmax of single-dose rosuvastatin | During administration of rosuvastatin (Treatment A) and both rosuvastatin and ACT-541468 (Treatment B2); i.e. for about 2 weeks.
  Effect of ACT-541468 at steady-state on tmax of single-dose rosuvastatin
Effect of ACT-541468 at steady-state on AUC0-t of single-dose rosuvastatin | During administration of rosuvastatin (Treatment A) and both rosuvastatin and ACT-541468 (Treatment B2); i.e. for about 2 weeks.
  Effect of ACT-541468 at steady-state on AUC0-t of single-dose rosuvastatin
Effect of ACT-541468 at steady-state on AUC0-∞ of single-dose rosuvastatin | During administration of rosuvastatin (Treatment A) and both rosuvastatin and ACT-541468 (Treatment B2); i.e. for about 2 weeks.
  Effect of ACT-541468 at steady-state on AUC0-∞ of single-dose rosuvastatin
Effect of ACT-541468 at steady-state on t½ of single-dose rosuvastatin | During administration of rosuvastatin (Treatment A) and both rosuvastatin and ACT-541468 (Treatment B2); i.e. for about 2 weeks.
  Effect of ACT-541468 at steady-state on t½ of single-dose rosuvastatin

SECONDARY OUTCOMES:
Trough concentration (Ctrough) of ACT-541468 | During ACT-541468 administration (Treatment B1 and B2); i.e. for about 1 week
  Trough concentration (Ctrough) of ACT-541468
Change in vital signs | From Screening to EOS (for a maximum of up to 5 weeks)
  Change from baseline to each time point of measurement during each treatment in vital signs (supine BP and pulse rate)
Change in ECG variables | From Screening to EOS (for a maximum of up to 5 weeks)
  Change from baseline to each time point of measurement during each treatment in ECG variables
Treatment-emergent (serious) adverse events | From Screening to EOS (for a maximum of up to 5 weeks)
  Treatment-emergent AEs and SAEs during each treatment
Treatment-emergent ECG abnormalities | From Screening to EOS (for a maximum of up to 5 weeks)
  Treatment-emergent ECG abnormalities during each treatment
Change in body weight | From Screening to EOS (for a maximum of up to 5 weeks)
  Change from baseline to each time point of measurement during each treatment in body weight
Change in clinical laboratory tests | From Screening to EOS (for a maximum of up to 5 weeks)
  Change from baseline to each time point of measurement during each treatment in clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Mühlan, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Cepha s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No